CLINICAL TRIAL: NCT01207726
Title: Randomized Phase II Trial of Adjuvant Combined Epigenetic Therapy With 5-Azacitidine and Entinostat in Resected Stage I Non-small Cell Lung Cancer Versus Standard Care
Brief Title: Azacitidine and Entinostat in Treating Patients With Stage I Non-Small Cell Lung Cancer That Has Been Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual due to patients not wanting daily clinic administration of 5AZA and/or 6 months of treatment after surgery.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02901; NCI-2012-02901 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA_00038631; J1037 (Other: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital); 8311 (Other: CTEP); P30CA006973 (NIH)
Record Dates: First submitted 2010-09-10; First posted 2010-09-23 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine; entinostat

ARMS (2):
- Arm I (azacitidine, entinostat) (Experimental): Patients receive azacitidine SC on days 1-5 and 8-10 and entinostat PO QD on days 3 and 10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Other: Laboratory Biomarker Analysis
- Arm II (standard of care) (No Intervention): Patients receive standard of care.

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm I (azacitidine, entinostat)
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
  Arms: Arm I (azacitidine, entinostat)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (azacitidine, entinostat)

SUMMARY:
This study combines the deoxyribonucleic acid (DNA) methyltransferase inhibitor, 5-azacitidine (5-AZA), with an orally bioavailable histone deacetylase inhibitor, entinostat (SNDX-275), for the adjuvant treatment of patients with resected stage I non-small cell lung cancer (NCSLC).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of 5-azacitidine and entinostat on the hazard of 3 year progression-free survival in patients with resected stage I non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. To assess the safety, tolerability and toxicity of entinostat and 5-azacitidine in patients with resected stage I non-small cell lung cancer.

II. To explore the effect of entinostat and 5-azacitidine on median disease-free and overall survival in patients with resected stage I non-small cell lung cancer.

III. To assess the pharmacodynamic effects of 5-azacitidine and entinostat on DNA methylation and gene re-expression in patients with resected stage I NSCLC through analysis of sputum.

IV. To estimate the effect of entinostat and 5-azacitidine on progression free survival comparing patients with N2 lymph nodes categorized as methylated pre-treatment with those who are categorized as unmethylated.

V. To establish factors that predict clinical outcome in patients treated with combination epigenetic therapy by performing genome-wide analyses on pre-treatment tumor DNA.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive azacitidine subcutaneously (SC) on days 1-5 and 8-10 and entinostat orally (PO) once daily (QD) on days 3 and 10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive standard of care.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be status post complete (R0) surgical resection of pathologically-proven NSCLC (stage IA-IB according to AJCC version 7)
* Patients must be at least 4 weeks out from completion of surgery
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal
* The effects of entinostat and 5-azacitidine on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients must be within 8 weeks of completing surgery
* Patients who have received prior chemotherapy or radiation for treatment of their current diagnosis of lung cancer
* Patients with sub-lobar resections (ie: wedge resection or segmentectomy)
* Patients without mediastinal lymph node specimens from mediastinoscopy or surgery (at least level R4 or 7 for right sided tumors OR at least level 5, 6 or 7 for left sided tumors)
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat, 5-azacitidine or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because entinostat and 5-azacitidine are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with entinostat or 5-azacitidine, breastfeeding should be discontinued if the mother is treated on this protocol; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with entinostat or 5-azacitidine; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital
Locations (9):
- United States (9):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Azacitidine SC and Entinostat Oral: Patients receive azacitidine SC on days 1-5 and 8-10 and entinostat PO QD on days 3 and 10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Chemotherapy Alone: Standard of care chemotherapy
Period: Overall Study
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Azacitidine SC and Entinostat PO: Patients receive azacitidine SC on days 1-5 and 8-10 and entinostat PO QD on days 3 and 10. Followed by Cytotoxic Therapy investigator Choice
- Cytotoxic Therapy: Standard of care
- Total: Total of all reporting groups
Arm/Group | Azacitidine SC and Entinostat PO | Cytotoxic Therapy | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants] — Population: Study stopped due to early stopping rule
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 4 | 1 | 5
    >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Full Range); unit: years] | 66 [58 to 70] | 68 [61 to 72] | 67 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: The DFS hazard rate and 95% confidence interval will be reported. At this time, event time distributions for disease-free survival in the two arms will be estimated with the method of Kaplan and Meier and compared using a stratified Cox-proportional hazards model (stratified for stage IA vs IB) with a two-sided alpha of 10%.
Time Frame: 3 years
Population: The study was terminated early due to poor accrual since the requirement of clinic administration of the 5AZA daily and post-operative patients not wanting 6 months of treatment. Data was not collected to assess this outcome measure.
Arm/Group | Arm I (Azacitidine, Entinostat) | Arm II (Standard of Care)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Factors That Predict Clinical Outcome in Patients Treated With Combination Epigenetic Therapy in Terms of Epigenomic Data Generated From the Illumina Platform
Description: The study was terminated early due to poor accrual since the requirement of clinic administration of the 5AZA daily and post-operative patients not wanting 6 months of treatment. For this reason, 13 pts were enrolled and data was not analyzed, for which we are unable to make any conclusions or report results.
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Median Disease-free Survival
Description: Determined by the method determined by Kaplan and Meier. Estimated with 95% confidence intervals. Cox proportional hazard modeling will be used for multivariate analysis.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Relapses and Deaths Per Total Time of Follow-up Comparing Patients With N2 Lymph Nodes in Terms of Methylated and Unmethylated
Description: Kaplan Meier curves will be used.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: as for outcome 3
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat PO | Cytotoxic Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Presence of Methylation Patterns
Description: McNemar's test will be used to compare the change in methylation after treatment in sputum.
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Toxicities Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
Description: Simple descriptive statistics will be utilized to display the data.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Azacitidine SC and Entinostat Oral | Chemotherapy Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Groups:
- Azacitidine SC and Entinostat PO: Patients receive azacitidine SC on days 1-5 and 8-10 and entinostat PO QD on days 3 and 10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Cytotoxic Chemotherapy: Investigators Choice Chemotherapy
Arm/Group | Azacitidine SC and Entinostat PO | Cytotoxic Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less